CLINICAL TRIAL: NCT05794035
Title: Impact of Hypofractionated Radiotherapy Strategy After Surgery of Skin Carcinomas in Older Patients IMPACTE-01
Brief Title: Impact of Hypofractionated Radiotherapy Strategy After Surgery of Skin Carcinomas in Older Patients
Acronym: IMPACTE-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP180682
Record Dates: First submitted 2023-02-15; First posted 2023-03-31 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Skin Cancer, Non-Melanoma
Keywords: Non Melanoma Skin Cancer; Adjuvant radiation therapy; older patient
MeSH Terms: conditions — Skin Neoplasms | interventions — Surgical Procedures, Operative; four-arm poly(ethylene oxide)-b-poly(2-(diethylamino)ethyl methacrylate)

STUDY DESIGN:
Intervention Model Description: After inclusion of patient aged ≥ 70 years with performance status OMS 0-3 who had completed surgery (R0) for SCC and BCC with at least one unfavorable prognostic factor, the patients will be randomized in 3 arms with stratification by center, time from surgery to wound healing and perineural invasion.
  * Arm A: Surgery alone
  * Arm B: Surgery + Moderate HF 45Gy in 15 fractions, 3 fractions per week over 5 weeks to the operative bed.
  * Arm C: Surgery + Extreme HF : 30Gy in 5 fractions of 6Gy, 1 fraction per week, over 5 weeks to the operative bed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Surgery alone (Active Comparator): After inclusion of patient aged ≥ 70 years with performance status OMS 0-3 who had completed surgery (R0) for SCC and BCC with at least one unfavorable prognostic factor, patient will have surgery alone with no hypo fractionation treatment
  Interventions: Other: Surgery alone, without radiation post surgery
- Surgery + Moderate hypo fractionation (HF) (Experimental): Surgery + Moderate hypo fractionation (HF) 45Gy in 15 fractions, 3 fractions per week over 5 weeks to the operative bed.
  Interventions: Other: Surgery with additional moderate hypofractionation RT (15 fractions)
- Surgery + Extreme hypo fractionation (HF) (Experimental): Surgery + Extreme hypo fractionation (HF): 30Gy in 5 fractions of 6Gy, 1 fraction per week, over 5 weeks to the operative bed.
  Interventions: Radiation: Surgery with extreme hypo fractionation treatment (HF)

INTERVENTIONS:
Other: Surgery with additional moderate hypofractionation RT (15 fractions) — After randomization, patients will then be followed-up at 3 months post randomization and at each surveillance visit (M6, M12, M24 and M36).
  Adjuvant Radiotherapy:
  -Arm B: Surgery followed by moderate hypofractionation RT (15 fractions): 45Gy in 15 fractions, 3 fractions per week over 5 weeks to the operative bed.
  Other Names: Arm B:
  Arms: Surgery + Moderate hypo fractionation (HF)
Other: Surgery alone, without radiation post surgery — Arm A: Surgery alone followed by surveillance
  Arms: Surgery alone
Radiation: Surgery with extreme hypo fractionation treatment (HF) — After randomization, patients will then be followed-up at 3 months post randomization and at each surveillance visit (M6, M12, M24 and M36).
  Adjuvant Radiotherapy:
  -Arm C= Surgery followed by extreme hypofractionation RT (5 fractions, 2 fractions/week): 30Gy in 5 fractions of 6Gy over 5 weeks to the operative bed.
  Other Names: Arm C
  Arms: Surgery + Extreme hypo fractionation (HF)

SUMMARY:
Non-melanoma skin cancer (NMSC) incidence as well as morbidity rates are high in older patients. Surgery is the standard of care. About 5 to 10% of NMSC present high-risk clinico-pathologic features that can increase risk of local recurrence (LR).

Adjuvant radiation therapy (ART) is often discussed regarding the risk of local recurrence. Despite the lack of high level evidence, ART is indicated in patients according to unfavorable prognostic factors. ART benefit is generally questioned in regard to the potential degradation of the patient's quality of life (QoL). Currently there is no prospective trial or recommendations that take into account geriatric patients' evaluation and profiles during the management of NMSC. In addition, there is no data that could help to define the subgroup of elderly patients who will benefit from ART in tumors with unfavorable prognostic factors.

In terms of ART, multiple fractionation schedules are available, ranging from standard fractionation (45-60Gy in 5-6 weeks) to the extreme hypofractionation (HF) delivering 16-18Gy in one fraction.

In routine practice, HF is mainly preferred in elderly patients for more convenience by reducing the number of transports and increase health related quality of life (HRQoL). However, there is no data on the fragility profiles of these patients, nor validating any HF schedule in terms of efficacy, acute toxicity, cosmetic results, and impact on HRQoL.

the main ain objective is to evaluate the comparative efficacy of two modalities of Radiotherapy over surgery alone on local tumor control in older patients with Non Melanoma Skin Cancer (NMSC) In current practice, adjuvant radiotherapy is discussed regarding the risk of local recurrence as determined by the existence (or not) of unfavorable prognostic factors. The proposed study will include R0-high risk of CBC and CEC of the skin in elderly patients. There is no risk regarding the design of the trial as the last will respond to two important unknown questions regarding the utility of RT and its fractionation in this population. Moreover, it is an excellent opportunity to collect prospectively geriatric evaluation and HRQoL data that are lacking in the literature for skin cancers. No constraints are seen neither in the design, nor in the potential recruitments.

DETAILED DESCRIPTION:
A short description, 5000 characters

Intro:

Non-melanoma skin cancer (NMSC) incidence as well as morbidity rates are high in older patients. Surgery is the standard of care. About 5 to 10% of NMSC present high-risk clinico-pathologic features that can increase risk of local recurrence (LR).

Adjuvant radiation therapy (ART) is often discussed regarding the risk of local recurrence. Despite the lack of high level evidence, ART is indicated in patients according to unfavorable prognostic factors. ART benefit is generally questioned in regard to the potential degradation of the patient's quality of life (QoL). Currently there is no prospective trial or recommendations that take into account geriatric patients' evaluation and profiles during the management of NMSC. In addition, there is no data that could help to define the subgroup of elderly patients who will benefit from ART in tumors with unfavorable prognostic factors.

In terms of ART, multiple fractionation schedules are available, ranging from standard fractionation (45-60Gy in 5-6 weeks) to the extreme hypofractionation (HF) delivering 16-18Gy in one fraction.

In routine practice, HF is mainly preferred in elderly patients for more convenience by reducing the number of transports and increase health related quality of life (HRQoL). However, there is no data on the fragility profiles of these patients, nor validating any HF schedule in terms of efficacy, acute toxicity, cosmetic results, and impact on HRQoL.

Hypothesis/Objective

Main Objective:

To evaluate the comparative efficacy of two modalities of Radiotherapy over surgery alone on local tumor control in older patients with Non Melanoma Skin Cancer (NMSC) In current practice, adjuvant radiotherapy is discussed regarding the risk of local recurrence as determined by the existence (or not) of unfavorable prognostic factors. The proposed study will include R0-high risk of CBC and CEC of the skin in elderly patients. There is no risk regarding the design of the trial as the last will respond to two important unknown questions regarding the utility of RT and its fractionation in this population. Moreover, it is an excellent opportunity to collect prospectively geriatric evaluation and HRQoL data that are lacking in the literature for skin cancers. No constraints are seen neither in the design, nor in the potential recruitments.

Primary endpoint:

Local tumor control at 3-year follow-up in a time-to-event analysis Method This is a multicenter, randomized, open-labeled, comparative 3 arms phase III trial.

After inclusion of patient aged ≥ 70 years with performance status OMS 0-3 who had completed surgery (R0) for SCC and BCC with at least one unfavorable prognostic factor, all patientsst will have G8 score and a Geriatric Core Data Set (G CODE) evaluation. Performance of a complete oncogeriatric evaluation and its modalities will be left to the discretion of the investigator.

The patients will be randomized in 3 arms with stratification by center, time from surgery to wound healing and perineural invasion.

* Arm A: Surgery alone
* Arm B: Surgery + Moderate HF 45Gy in 15 fractions, 3 fractions per week over 5 weeks to the operative bed.
* Arm C: Surgery + Extreme HF : 30Gy in 5 fractions of 6Gy, 1 fraction per week, over 5 weeks to the operative bed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 70 years
* OMS 0-3
* Pathology confirmation of invasive SCC or BCC
* At least one of high-risk factors for recurrence (R0 but close margins, location/size, microscopic perineural invasion, recurrent primary disease, immunosuppression, thickness including Breslow and Clark level, poorly-moderately differentiated)
* No indication of regional nodal RT
* No prior RT to the treated site
* Written consent from patient or his/her legal representative, trustworthy person or family member if the person is physically unable to give his or her written consent
* Life expectancy ≥ 6 months, as clinically estimated by the investigator in charge of enrolment
* No contraindication for surgery and RT after multidisciplinary board meeting evaluation
* Affiliated to a social security scheme

Exclusion Criteria:

* Macroscopic incomplete resection of the primary tumor (≥ R1)
* Patient with severe dementia not allowing follow-up
* Any psychological, familial, sociological, geographical or logistical reasons that would prevent participation to surveillance during treatment and follow-up
* Other active cancers in treatment
* Participation in another interventional study (therapeutic trial interfering with the study's endpoints)
* Patient on AME (state medical aid)
* Persons deprived of their liberty by a judicial or administrative decision

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 303 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | at 3 years
  Levels and changes from baseline in HRQoL as assessed by the cancer-specific European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) and QLQ-ELD14 module developed for older patients with cancer, and treatment burden, as assessed by an adapted version of the Treatment Burden Questionnaire (TBQ; EVALUATION AT
QLQ-ELD14 Questionnaire | at 3 years
  Levels and changes from baseline in HRQoL as assessed by the cancer-specific European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) and QLQ-ELD14 module developed for older patients with cancer, and treatment burden, as assessed by an adapted version of the Treatment Burden Questionnaire (TBQ; EVALUATION AT
rate of Toxicity | during RadiotherapyT
  Acute and late toxicity, as assessed by CTCAE v4.03 criteria
efficacy of treatment modalities on regional recurrence (RR), at 3-year follow-up | at 3 years
progression-free survival (PFS) | at 3-year follow-up
overall survival (OS) | at 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No